CLINICAL TRIAL: NCT02124590
Title: The Effect of Oral Carnitine Supplementation on MRS-derived Mitochondrial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053117
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Elderly; Pre-diabetic
Keywords: Carnitine; Acylcarnitine; Exercise; Exercise Intensity; Insulin Sensitivity
MeSH Terms: conditions — Glucose Intolerance; Motor Activity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute Exercise (Experimental): Repeated isometric leg exercises at varying intensities and a second visit with aerobic bike exercise for 30 minutes at 50% peak VO2.
  Interventions: Other: Acute Exercise

INTERVENTIONS:
Other: Acute Exercise — Repeated isometric leg exercises at varying intensities for up to twelve minutes per bout. Leg exercises will target the quadriceps muscles.
Other: Acute Exercise — Aerobic exercise session on a bike at 50% of peak VO2 for 30 minutes.

SUMMARY:
This is a longitudinal study supported by Pfizer and is a collaboration between DMPI (Duke Molecular Physiology Institute) and DIAL (Duke Image Acquisition Laboratory) to measure the effects of acute exercise on carnitine and acylcarnitine levels in the muscle and on insulin sensitivity in the plasma. This pilot study seeks to explain why moderate intensity exercise provides more improvements in glucose control for pre-diabetic patients than vigorous intensity. The investigators hypothesize that moderate intensity exercise might be beneficial for elderly individuals who are overweight or obese, specifically by: 1. Reducing damaging excess protein acetylation (measured in muscle biopsy), 2. Improving the acylcarnitine/carnitine ratio (measured by MRS), 3. Improving overall mitochondrial function as reflected in reduced phosphocreatine recovery time (measured by MRS) and 4. Increasing insulin sensitivity as measured by a 4-hour oral glucose tolerance test. Investigators intend to use the results of this study to show feasibility in measuring mitochondrial function at Duke for a larger federal grant submission. Investigators hypothesize that carnitine insufficiency might contribute to mitochondrial dysfunction and obesity-related impairments in glucose tolerance and insulin action.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60-80 years
* Moderately Overweight: BMI - 25.0 - 35.4
* Sedentary - exercise ≤ 1 day/week
* Fasting plasma glucose: > 100 - < 126 mg/dL
* Readings from two separate days

Exclusion Criteria:

* Orthopedic limitations, musculoskeletal disease and/or injury
* Allergic to xylocaine
* Inability to give blood continuously through an intravenous catheter
* Have a confounding medical condition that is progressive and unstable such as HIV, Hepatitis C, active cancer, and/or taking medications for those conditions that are likely to confound the assessment of pre-diabetes
* Prior surgical operation within the past 6 months
* Prior injury to the eye involving metallic objects or fragments
* Prior injury involving a metallic object or foreign body (eg. BB, bullet, shrapnel, etc.)
* Tattoos from the waist down to the feet
* Any of the following implants or devices

  * Aneurysm clip
  * Cardiac pacemaker
  * Implanted cardioverter defibrillator (ICD)
  * Electronic implant or device
  * Magnetically activated implant or device
  * Neurostimulation system
  * Spinal cord stimulator
  * Internal electrodes or wires
  * Bone growth/bone fusion stimulator
  * Cochlear, otologic or other ear implant
  * Insulin or other infusion pump
  * Implanted drug infusion device
  * Eye implants
  * Vascular access port and/or catheter
  * Wire mesh implant or stent
  * Other implant
* Claustrophobia
* Prior knee replacement surgery
* Pregnant or intending to become pregnant during the study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Acylcarnitine/Carnitine ratio | Baseline, One Month

SECONDARY OUTCOMES:
Change in Protein acetylation | Baseline, One Month
Change in Insulin Sensitivity | Baseline, One Month
Change in Mitochondrial Function | Baseline, One Month

CONTACTS AND LOCATIONS:
Overall Officials: William E Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States